CLINICAL TRIAL: NCT06984718
Title: A Phase II, Randomized, Open-label, Multi-center Study of AK104 in Combination With Lenvatinib Versus Lenvatinib in Patients With Advanced Hepatocellular Carcinoma Who Have Progressed on Atezolizumab and Bevacizumab
Brief Title: A Phase II Study of AK104 Combination With Lenvatinib Versus Lenvatinib for Second-line HCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-225
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: HCC; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AK104+lenvatinib (Experimental): AK104 IV plus lenvatinib orally
  Interventions: Biological: AK104+lenvatinib
- lenvatinib (Active Comparator): lenvatinib orally
  Interventions: Drug: lenvatinib

INTERVENTIONS:
Biological: AK104+lenvatinib — Subjects will receive AK104+lenvatinib until disease progression
  Arms: AK104+lenvatinib
Drug: lenvatinib — Subjects will receive lenvatinib until disease progression
  Arms: lenvatinib

SUMMARY:
This is a Phase II, randomized, open-label, global, multi-center study to compare the efficacy and safety of AK104 in combination with lenvatinib versus lenvatinib in patients with advanced hepatocellular carcinoma who have progressed on the first line treatment of atezolizumab and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the Informed Consent Form (ICF) voluntarily.
2. Age ≥18 years at time of signing ICF.
3. Histologic or cytologic confirmation of HCC, or clinical diagnosis of HCC as per AASLD criteria.
4. BCLC stage B or C, and not suitable for curative surgical or local therapy.
5. Participants have progressed on the prior first-line systemic treatment with atezolizumab plus bevacizumab combination treatment.
6. At least one measurable lesion according to RECIST v1.1.
7. Child-Pugh Class A .
8. ECOG performance status of 0 or 1.
9. With a life expectancy of ≥3 months.
10. Adequate organ and hematologic function.

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
2. Tumor thrombus invasion of superior mesenteric vein.
3. Has a known history of, or any evidence of CNS metastases.
4. Has received anti-cancer therapy for HCC within 3 weeks prior to the first dose of study treatment.
5. Has received systemic anti-cancer therapy other than atezolizumab and bevacizumab.
6. Has participated in another clinical study within 4 weeks prior to the first dose.
7. History of liver transplantation.
8. History of hepatic encephalopathy.
9. Clinically symptomatic or recurrently drained pleural effusion, pericardial effusion, or ascites.
10. History of bleeding event due to esophageal and/or gastric varices within 6 months prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST v1.1 by Blinded Independent Central Review (BICR) | Up to 24 months
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by BICR according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from randomization to death due to any cause.
Progression-free survival (PFS) assessed by investigator per RECIST v1.1 | Up to 24 months
  PFS is defined as the time from randomization till the first documented disease progression (Per RECIST v1.1 assessed by the investigator) or death due to any cause, whichever occurs first.
Duration of Response (DOR) assessed by investigator per RECIST v1.1 | Up to 24 months
  DOR means time measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Time to Response (TTR) assessed by investigator per RECIST v1.1 | Up to 24 months
  TTR refers to Time to Response.
Number of participants with adverse event (AE) | Up to 24 months
  The number of participants experiencing an Adverse Event (AE) and the severity of AEs will be assessed. AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Finn, Ph.D., Principal Investigator — Department of Medicine, University of California; Jian Zhou, Ph.D., Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No